CLINICAL TRIAL: NCT04872881
Title: Comparison of Effectiveness of Different Airway Management Methods During Fiberoptic Bronchoscopy Assisted Percutaneous Tracheostomy
Brief Title: Comparison of Effectiveness of Different Airway Management Methods During Percutaneous Tracheostomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Elif Göktaş, Anesthesiology Resident, Bozyaka Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: eliftez
Record Dates: First submitted 2021-04-22; First posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Intubation, Intratracheal; Tracheostomy; Laryngeal Masks; Intensive Care Units
Keywords: Percutan Dilatational Tracheostomy; Intensive Care Units
MeSH Terms: interventions — Intubation, Intratracheal; Propofol; Rocuronium; Fentanyl

STUDY DESIGN:
Intervention Model Description: There are two groups: ETT Group and LMA Group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ETT Group (Active Comparator): ETT will be repositioned with direct laryngoscopy (ETT cuff will be inflated just above the vocal cords). "The Reposition Time" will start with the cuff deflation and end with successful ventilation after repositioning. If the ETT can not be repositioned within 5 minutes, it will be considered as a "Failed Airway" and tracheostomy will be continued with the usual method (ETT cuff will be inflated under the vocal cords)
  Interventions: Procedure: Endotracheal Tube Insertion; Procedure: Fiberoptic Bronchoscopy; Procedure: Radial Artery Monitoring; Diagnostic Test: Anteroposterior chest x-ray; Diagnostic Test: Arterial Blood Gas Analyses; Drug: Propofol Fresenius; Drug: Rocuronium; Drug: Fentanyl
- LMA Group (Active Comparator): After selecting the appropriate LMA size for the patient, the ET Tube will be removed and the LMA will be inserted. "The LMA Insertion Time" will start with the cuff deflation of the ETT and end with successful ventilation after LMA insertion. If the LMA cannot be inserted in 3 attempts, it will be considered as a "Failed Airway" and tracheostomy will be continued with the usual method (ETT cuff will be inflated under the vocal cords)
  Interventions: Procedure: Laryngeal Mask Insertion; Procedure: Fiberoptic Bronchoscopy; Procedure: Radial Artery Monitoring; Diagnostic Test: Anteroposterior chest x-ray; Diagnostic Test: Arterial Blood Gas Analyses; Drug: Propofol Fresenius; Drug: Rocuronium; Drug: Fentanyl

INTERVENTIONS:
Procedure: Endotracheal Tube Insertion — ETT will be repositioned with direct laryngoscopy (ETT cuff will be inflated just above the vocal cords)
  Arms: ETT Group
Procedure: Laryngeal Mask Insertion — After selecting the appropriate LMA size for the patient, the ET Tube will be removed and the LMA will be inserted.
  Arms: LMA Group
Procedure: Fiberoptic Bronchoscopy — After the patients' airway is established, the trachea and the process area will be displayed by the physician.
  The success rate will be increased by performing the procedure with fiberoptic bronchoscopy.
Procedure: Radial Artery Monitoring — The radial artery will be cannulated. Hemodynamic monitoring and blood gas analysis will be done in this way.
Diagnostic Test: Anteroposterior chest x-ray — When the tracheostomy cannula is placed and the patient is ventilated, the procedure will be terminated and confirmed with anteroposterior chest x-ray.
Diagnostic Test: Arterial Blood Gas Analyses — Hypoxia, acidosis and carbon dioxide increase will be followed
Drug: Propofol Fresenius — 2mg/kg of propofol 2% injectable solution was given and propofol infusion at the dose of 6 mg/kg/hour will be started.
Drug: Rocuronium — 0.6 mg/kg of rocuronium 50mg/5ml injectable solution was given.
  Other Names: Muscuron
Drug: Fentanyl — 1mcg/kg fentanyl of 0.5 mg/10ml injectable solution was given.

SUMMARY:
Tracheostomy is a vital procedure in the ICU to maintain the airway and prevent complications that may occur due to intubation. It helps reduce the dead space volume, airway resistance and provides comfort to the patients during the weaning from mechanical ventilation. Two methods are widely used in Percutaneous Dilatational Tracheostomy (PDT): The multiple dilation method (Ciaglia) and the Griggs method.Griggs method will be used in the study.

The Griggs Method: A 10-15 millimeter skin incision is made between the level of the second-third tracheal rings. The location of the needle is confirmed by entering the trachea with an injector filled with 2-3 mL saline from the midline and aspirating air. A J-tipped guidewire is advanced through the needle and the needle is removed. A special forceps with a channel at the tip, through which the guidewire can pass is used in this method. The forceps advanced through the guidewire and then subcutaneous tissues and trachea are dilated in one or two steps. When the stoma is large enough to insert the cannula, it is placed in the trachea and fixed.

Patients who will undergo tracheostomy in the ICU will be included in the study and randomly assigned into two groups. Two different methods, endotracheal tube (ET) or laryngeal mask (LMA), will be used during the tracheostomy for airway management. In both methods, fiberoptic bronchoscopy will assist the procedure.

Researchers aim to compare the two airway management methods in terms of complications, procedure time, and the number of staff needed.

DETAILED DESCRIPTION:
Protection of the airway during percutaneous tracheostomy can be achieved with an endotracheal tube (ETT) or laryngeal mask (LMA).Researchers aimed to compare the use of ETT and LMA in this prospective, randomized study.

Multiple blood gas analyses will be performed during the procedure. Airway failure rates, total procedure time, the occurrence of gastric distension and regurgitation, number of staff needed, complications (Hypercarbia, hypoxia, etc.), and hemodynamic parameters (Non-invasive blood pressure, pulse oximeter, electrocardiogram) will be compared.

Patients will be divided into two groups with simple randomization. A-priori study with 14 patients suggested 52 patients are needed for statistical significance (G*Power 3.1 software was used). Patients will be reviewed for suitability for procedure as stated in the inclusion criteria. Patients and/or relatives will be informed about the study and informed consent will be obtained. Invasive arterial blood pressure monitoring of the patients will be available. Before the procedure, the patients' fasting period for 6 hours will be completed and the nasogastric catheter will be removed. Arterial blood gas sample will be checked before the procedure begins. By placing a transverse elevation under the shoulders, the patients' neck will be extended as appropriate. Patients will be positioned after induction with 2 mg/kg propofol, 0.6 mg/kg rocuronium, and 1 mcg/kg fentanyl IV, and positioning time will be recorded. Propofol infusion at the dose of 6 mg/kg/hour will be started. Electrocautery will be available. Patients will be mechanically ventilated with a controlled mode (CMV) with 7ml/kg tidal volume, 15/min frequency, and 5 cmH2O PEEP. Preoxygenation will be made with 100% FiO2 for 5 minutes.

ETT Group: ETT will be repositioned with direct laryngoscopy (ETT cuff will be inflated just above the vocal cords). "The Reposition Time" will start with the cuff deflation and end with successful ventilation after repositioning. If the ETT can not be repositioned within 5 minutes, it will be considered as a "Failed Airway" and tracheostomy will be continued with the usual method (ETT cuff will be inflated under the vocal cords).

LMA Group: After selecting the appropriate LMA size for the patient, the ET Tube will be removed and the LMA will be inserted. "The LMA Insertion Time" will start with the cuff deflation of the ETT and end with successful ventilation after LMA insertion. If the LMA cannot be inserted in 3 attempts, it will be considered as a "Failed Airway" and tracheostomy will be continued with the usual method (ETT cuff will be inflated under the vocal cords).

After the ventilation is provided, arterial blood gas samples will be analyzed at the 3rd, 6th, and 10th minutes and every 5 minutes afterward until the end of the procedure. In both groups, fiberoptic bronchoscopy will assist the procedure and "Duration of the Confirmation of the Incision Site" will be noted. The bronchoscopy period will start when the physician who will perform the bronchoscope takes the bronchoscope in his hand and ends with the confirmation of the incision site. The area will be cleaned with iodide skin antiseptic, covered with a sterile cover, and surgical tools and tracheostomy kit will be prepared for the procedure. This will be recorded as "Preparation Time". Tracheostomy will preferably be performed between the 2nd and 3rd cartilage rings but one upper or lower level will be used if needed (per patients' anatomy). Local anesthesia will be applied for the incision site with 4 ml of local anesthetic solution containing %2 lidocaine and %0,00125 epinephrine. "Procedure Time" will start with skin incision and end with successful ventilation after the tracheostomy cannula cuff is inflated.

Gastric distension, hypoxia, regurgitation, hemodynamic parameters (every 3 minutes), complications, and the number of staff will be recorded. When the tracheostomy cannula is placed and the patient is ventilated, the procedure will be terminated and confirmed with an anteroposterior chest x-ray.

SPSS (Statistical Package for Social Sciences version 24) was used for statistical calculation. Parametric test results were reported as mean and standard deviation and non-parametric test results as number and percentage or median and interquartile range. The compliance of the data to normal distribution was determined by the single sample Kolmogorov-Smirnov test. Normally distributed quantitative data were compared with the independent sample T-Test, quantitative data that did not follow normal distribution were compared with the Mann-Whitney U test. A Chi-square test was used to compare qualitative data.

The significance level was determined as p <0.05 at the 95% confidence interval for the analyzes.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant patients over 18 years of age
* Patients who need a tracheostomy
* Patients whose opening method of tracheostomy is suitable for percutaneous tracheostomy.

Exclusion Criteria:

* Refusal of the procedure by the patient or her legal representative
* Patients under the age of 18
* Body mass index> 35 patient group
* Patients with a mass in the neck region for any reason
* Skin infection at the procedure site
* Coagulopathy
* Inability to palpate the cricoid cartilage

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Arterial Blood Gas Analysis | Before the procedure
  Monitoring of hypoxia, acidosis, and carbon dioxide
Arterial Blood Gas Analysis | 3rd minute after ventilation
  Monitoring of hypoxia, acidosis, and carbon dioxide
Arterial Blood Gas Analysis | 6th minute after ventilation
  Monitoring of hypoxia, acidosis, and carbon dioxide
Arterial Blood Gas Analysis | 10th minute after ventilation
  Monitoring of hypoxia, acidosis, and carbon dioxide
Arterial Blood Gas Analysis | When the tracheostomy cannula cuff is inflated
  Monitoring of hypoxia, acidosis, and carbon dioxide
Positioning time | Before the procedure
  By placing a transverse elevation under the shoulders, the patients' neck will be extended as approprite.
The Reposition Time | Before the procedure
  The Reposition Time will start with the cuff deflation and end with successful ventilation after repositioning. If the ETT can not be repositioned within 5 minutes, it will be considered as a "Failed Airway".
The LMA Insertion Time | Before the procedure
  The LMA Insertion Time will start with the cuff deflation of the ETT and end with successful ventilation after LMA insertion. If the LMA cannot be inserted in 3 attempts, it will be considered as a "Failed Airway"
Duration of the Confirmation of the Incision Site | Before the procedure
  The bronchoscopy period will start when the physician who will perform the bronchoscope takes the bronchoscope in his hand and ends with the confirmation of the incision site
Preparation Time | Before the procedure
  Area will be cleaned with iodide skin antiseptic, covered with a sterile cover and surgical tools and tracheostomy kit will be prepared for the procedure
Procedure Time | 15 minutes after the procedure begins
  "Procedure Time" will start with skin incision and end with successful ventilation after tracheostomy cannula cuff is inflated.

SECONDARY OUTCOMES:
Incidence of gastric distension | Throughout the tracheostomy procedure
Incidence of hypoxia | Throughout the tracheostomy procedure
Incidence of regurgitation | Throughout the tracheostomy procedure
The number of staff needed | Throughout the tracheostomy procedure
Heart rate | Every 3 minutes during the procedure
Blood pressure | Every 3 minutes during the procedure
Pulse oximeter | Every 3 minutes during the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Elif Göktaş, Study Chair — Izmir Bozyaka Research and Trainings Hospital; Zeki T TEKGUL, Study Chair — Izmir Bozyaka Research and Trainings Hospital; Hüseyin ÖZKARAKAŞ, Study Chair — Izmir Bozyaka Research and Trainings Hospital

REFERENCES:
- See also: Laryngeal mask airway vs endotracheal tube to facilitate bedside percutaneous tracheostomy in critically ill patients: a prospective comparative study. — https://www.jpgmonline.com/article.asp?issn=0022-3859;year=2002;volume=48;issue=1;spage=11;epage=5;aulast=Ambesh
- See also: Laryngeal Mask Airway or Endotracheal Tube for Percutaneous Dilatational Tracheostomy — https://www.researchgate.net/publication/42806625_Laryngeal_Mask_Airway_or_Endotracheal_Tube_for_Percutaneous_Dilatational_Tracheostomy